# NEW YORK STATE PSYCHIATRIC INSTITUTE A STUDY OF L-DOPA FOR DEPRESSION AND SLOWING IN OLDER ADULTS

### Overview

Below is a summary of the study in which you are asked to participate. This outline is meant to be a guide for you to use while considering the study and reading the consent form. It is not meant to replace the consent form, which you will have to sign if you decide to participate in the study.

## Participation is Voluntary

As with all research, this is a voluntary study, and you do not have to participate if you do not want to. Also, you may stop participating at any time

### Alternatives

You do not have to participate in this study to receive treatment for depression or slowed thinking and movement. Antidepressant medication and psychotherapy are available outside of this study to treat depression. Exercise programs and cognitive remediation may be helpful for slowed thinking and movement and also are available outside this research project.

### Procedures

- At the beginning of the study, you will be given a physical examination, an electrocardiogram (EKG), and have your blood drawn.
  - Next you will have psychological tests and a test of your walking speed.
- One half of subjects in this study will undergo two (2) magnetic resonance imaging (MRI) scans of the brain and two (2) positron emission tomography (PET) scans of the brain. You may be offered participation in the treatment portion of the study if you are not eligible or do not wish to have MRI and PET scans.
- MRI scans use strong magnetic fields and radio waves to take pictures of your brain.
- The PET scans require placement of an IV catheter and injection of a radioactive substance called [11C]-raclopride. [11C]-raclopride allows us to examine a specific dopamine receptor in the brain which is important in some psychiatric diseases such as depression.
- All participants will receive treatment with a medication called carbidopa/levodopa (Sinemet) for 3 weeks.
- You will be asked to return each week to see one of the study doctors, talk about how you are feeling, and have tests of your thinking and walking speed.
- The research study will end after 3 weeks. You will fill out some psychological tests and have your thinking and walking speed tested again.



# Risks

This study includes some risks and discomforts (please refer to the consent form for further details and explanations of these risks). These include side effects associated with carbidopa/levodopa (such as nausea, headache, abnormal movements of arms and legs, muscle stiffness, and vivid dreams) and radiation exposure from the [11C]-raclopride tracer used in the PET scans.

# **Benefits**

This research study is not meant to benefit you directly. You may contact the study doctor, Dr. Bret Rutherford at 646-774-8660 with any questions.

#### PURPOSE OF STUDY

In this research study, you will receive a medication called carbidopa/levodopa (Sinemet). This medication is approved by the Food and Drug Administration for the treatment of Parkinson's Disease. We are using carbidopa/levodopa off-label in this study to see whether it is capable of improving depressive symptoms as well as mental and physical slowing that occur as people age.

In this study you may also be offered brain scans using magnetic resonance imaging (MRI) and positron emission tomorgraphy (PET). We are performing these scans to understand more about how Sinemet works in the brain. The PET scan involves the use of a radioactive investigational drug called [\$^{11}C\$]-raclopride. It is an investigational drug that attaches to parts of your brain that process dopamine. The drug contains a very small radioactive tracer that can be "seen" by the PET camera. The PET camera then takes "pictures" of the chemical activity in the brain by detecting the radioactive signal of [\$^{11}C\$]-raclopride. You will also be asked to take the drug carbidopa/levodopa so that the PET techniques can measure the impact of this drug on the dopamine system in the brain.

This study is supported by a grant from the National Institute of Mental Health.

### **VOLUNTARY**

Participation in this study is voluntary. If you do not wish to participate in this study or decide to discontinue your participation in this study later, you will not lose any benefits to which you are otherwise entitled, including current or future treatment at New York State Psychiatric Institute or Columbia University Medical Center. We will notify you of any significant new findings that may relate to your willingness to continue to participate.

### ALTERNATIVE TREATMENT

You do not have to participate in this study. The alternative to participating in this study is to seek treatment outside the research project so that you would be certain of receiving a medication approved for treatment of depression. Approved medications for depression are available (e.g., fluoxetine (Prozac), sertaline (Zoloft), etc), and psychotherapy also may be helpful with depression, whether on its own or combined with medication.

Although no treatments for mental and physical slowing have been formally approved by the FDA, other treatment approaches included exercise programs and cognitive training.

Information being collected is for research purposes only and is to learn more about changes in the brain's dopamine system with aging, not about you. It is not necessary to participate in this research study to have an MRI, and the MRI done as part of this study is not the same as one done for medical purposes.

### **STUDY PROCEDURES**

<u>Evaluation</u>: If you decide to participate in this study, you will have blood drawn, complete some psychological tests, and have your walking speed measured. The total amount of blood taken at this study visit is about two tablespoons. Results of these blood tests will be available to you, should you request them. The psychological tests measure thought processes such as memory, language, reasoning, and attention. These tests are paper-and-pencil and take about one hour to complete. The results of these tests are for research purposes only and will not be shared with you.

Based on these tests, it will be determined whether you are eligible for the treatment portion of the study. If you are not eligible, you will be referred to appropriate options for further treatment. If you are eligible and continue to wish to participate, you will proceed with the next part of the study.

MRI scans: Half of the participants in this study will be offered participation in brain imaging procedures. If you are otherwise eligible, you may participate in the treatment portion of the study if you are not eligible or do not wish to have MRI and PET scans. If you have brain imaging performed, you will have an MRI scan at the beginning of the study (before you receive any carbidopa/levodopa) and again at the end of the study (after you have taken carbidopa/levodopa for three weeks). The MRI uses strong magnetic fields and radio waves to take pictures of your brain. MRI involves lying on a table that slides into a large magnet shaped like a cylinder. Before beginning the imaging procedure, we will determine whether you have a pacemaker or any unsafe metallic implants such as an aneurysm clip or heart valve and certain tattoos, and you will be asked to remove any metal or magnetized objects (such as keys, chains, jewelry, retainers, medication patches, hairpins and credit cards). You will be asked to lie flat on your back in the MRI scanner for about 60 minutes and to remain as still as possible. You will not feel anything, but you will hear a knocking noise. This is a normal sound produced by the MRI scanner and does not indicate that anything is wrong.

<u>PET scans</u>: Individuals having brain imaging will also receive two PET scans, one at the beginning of the study (before you receive any carbidopa/levodopa) and again at the end of the study (after you have taken carbidopa/levodopa for three weeks). On the PET scan day, we will ask you not to eat from 6 am until the study is over. We will also ask you not to drink caffeinated beverages, such as coffee, tea, and soda, that day.

For the PET scans, we will need to place an intravenous catheter in one of your veins, and we will inject the radioactive substance through it. After the catheter is inserted, we will begin the PET scan. For both scans, we will ask you to lie on the narrow table. We will also position your head with a chin strap or a polyurethane headholder that we will mold around your head to reduce head movement during the scan. Right before each PET scan we will perform a very short (~10-15 second) CT scan of the brain which helps us make sure the PET scan is positioned correctly. We will then inject the radioactive substance [\$^{11}C\$]-raclopride through the catheter in your arm.

Each scan will last up to 1 hour. In addition, if you move your head during the PET scan we may do an additional CT position scan at the end of the PET scan. The second PET scan performed at the end of the study (three weeks after the first PET scan) will be done identical to the first scan. However, approximately 90 minutes before we give the second [\frac{11}{C}]-raclopride dose, we will ask you to take carbidopa/levodopa by mouth. After the end of the last scan, we will remove the catheter and you will be evaluated.

<u>Treatment study:</u> All participants (those who do the MRI, CT, and PET scans and those who do not) will then begin the starting dose of carbidopa/levodopa (37.5mg/150mg). This dose will be increased over the course of approximately 3 weeks to the final dose of 112.5mg/450mg. This will involve taking 4.5 pills per day, 1.5 in the morning, 1.5 at lunchtime, and 1.5 at night. You will receive free medication for the duration of the study.

If you have trouble tolerating the medication, we will lower your dose to one you previously tolerated. If you cannot tolerate any dose of the medication, your participation in the study will be discontinued. If the study doctor feels your condition worsens significantly, the current treatment will be stopped, and you will be offered different treatments for your slowed thinking and walking.

The study doctor may stop your participation in the study at any time without your consent if you do not comply with the study procedures or for other reasons. You will return each week to speak with the study doctor and have some tests. These appointments will last about 45 minutes. The research study will end after 3 weeks. During this week 3 visit, you will again fill out some psychological tests and have your walking speed measured.

Following the study, you will still receive 3 months of free doctor visits in the clinic. The medication used in this study is available from pharmacies, so it is an option to continue taking the medication following the study if you feel you have benefited from it. You will receive at least 1 month of free medication if you wish. Every effort will be made to provide free medication for 3 months total, but we cannot guarantee the

availability of free medication beyond 1 month. If you do not wish to continue the medication after the study, the dose will be gradually decreased over 3 days before stopping it.

### **RISKS**

<u>MRI risks:</u> While there have been no reports of any harmful long-term effects caused by 3T magnets or magnets of even higher strength, the long-term effects of being placed in a magnet of this strength are unknown. Also, although there are no known risks associated with pregnancy, we will not scan someone who is pregnant. If you are a female in your childbearing years, you will be asked to take a pregnancy test to ensure that you are not pregnant.

Some people have reported sensations during MRI scans with the 3T magnet, such as "tingling" or "twitching" (or, very rarely, a painful sensation), which are caused by changes in the magnetic field that can stimulate nerves in your body. With any MRI scan, on occasion, some people experience nervousness or discomfort due to the scanner's small space and the need to lie still. Except for pacemakers, some types of metallic implants, and medication patches, we are not aware of any other potentially dangerous interactions or hazards associated with the MRI scan. The MRI scanner also produces a loud noise; earplugs will be provided to reduce this discomfort. If you experience any discomfort and wish to stop the scan, you can tell the MRI technologist, and he or she will stop the scan immediately. In our experience, no one has had sensations from the MRI that did not stop when the scanning stopped.

<u>PET risks:</u> This research study involves exposure to radiation from Positron Emission Tomography (PET). Please note that this radiation exposure is not necessary for your medical care and is for research purposes only. The radiation you will receive in this study is from two [11C]-raclopride scans and from CT transmission scans of your head used to help obtain the PET images.

Everyone is exposed to natural background radiation daily from sources such as radon, food, water and the sun's rays. The average exposure of people in the U.S. each year is estimated to be 360 mrem (units for measuring radiation). As a very rough comparison, the amount of radiation you will receive in one PET scan is in the same range as what you would receive in one year from natural background sources. The amount of radiation you will receive in one CT scan is in the same range as what you would receive in 8 months from natural background sources. There are no known risks associated with receiving this level of radiation, however, radiation adds up throughout a person's lifetime. It is not possible to tell whether the small additional radiation received by participating in this study will increase your long-term risk for diseases such as cancer.

Please tell your study doctor or other study personnel if you have taken part in other research studies at NYSPI or other places/hospitals that used radiation. This way we can make sure that you will not receive too much radiation. You should consider x-rays taken in radiology departments, cardiac catheterization, and fluoroscopy as well as nuclear medicine scans in which radioactive materials were injected into your body. Before you take part in any future studies that use radiation, you should also tell those study doctors about your participation in this study.

Carbidopa/levodopa risks: The most common side effects reported for carbidopa/levodopa are nausea, headache, and vivid dreams. Patients who take carbidopa/levodopa for long periods of time to help with their Parkinson's Disease may experience the development of abnormal movements of their arms and legs, muscle stiffness, blood pressure changes, decreased appetite, and a wearing off effect of the medication. We do not expect these side effects will be applicable to you if you do not take the medication for more than several months. You should be careful about drinking alcohol, since it may have a greater effect on you in combination with medication.

*Other risks:* When your blood is drawn, there is a small risk you may be left with a bruise that will resolve within a few days. Results of blood tests taken for research purposes will remain confidential.

### **BENEFITS**

You may not benefit from this study, and no benefit is in any way guaranteed as a result of your participation.

### RESULTS OF YOUR MRI

While MRI scans are sometimes done for clinical purposes, the kind of MRI scan you may have as part of this study is for research purposes only. This means that the scans are not designed to provide clinical information that might be helpful to you or your doctor and they may not show problems that would normally be found in an MRI ordered to evaluate a specific medical problem. It is likely that the MRI scan will not have the quality of those done for clinical purposes.

However, within a month of the MRI scans, the scans will be read by a neuroradiologist for evidence of any obvious irregularities requiring your follow-up. You, or a physician whom you may designate, will be informed only when significant abnormalities are detected. If you wish, we can also inform you if there were no obvious findings. Given the nature of the scans, the absence of a finding does not mean that one is not present.

### CONFIDENTIALITY

Your records will be stored in a locked file and will only be available to the research staff and institutional personnel as part of routine audits. Representatives of the state and institutional regulatory personnel may review your records to ensure compliance with study design. There are legal advocacy organizations that have the authority under State Law to access otherwise confidential records, though they cannot be redisclosed without your consent. All records will be kept confidential to the extent permitted by law. Your name and other personal identifying information will be stored in an electronically secure database at New York State Psychiatric Institute. Electronically stored data will be accessible only by password known to the study investigators and research assistants. The results of your MRI scan also will be maintained in an electronically secure database at NYSPI and accessible only to the members of the research team.

Data from this study may be submitted to the National Institute of Mental Health Data Archive (NDA). NDA is a data repository run by the National Institute of Mental Health (NIMH) that allows researchers studying mental illness to collect and share deidentified information with each other. A data repository is a large database where information from many studies is stored and managed. De-identified information means that all personal information about research participants such as name, address, and phone number is removed and replaced with a code number. With an easier way to share, researchers hope to learn new and important things about mental illnesses more quickly than before.

During and after the study, the researchers will send de-identified information about your health and behavior to NDA. Other researchers nationwide can then file an application with the NIMH to obtain access to your de-identified study data for research purposes. Experts at the NIMH who know how to protect health and science information will look at every request carefully to minimize risks to your privacy.

You may not benefit directly from allowing your information to be shared with NDA. The information provided to NDA may help researchers around the world treat future children and adults with mental illnesses so that they have better outcomes. NIMH will also report to Congress and on its web site about the different studies that researchers are conducting using NDA data. However, you will not be contacted directly about the data you contributed to NDA.

You may decide now or later that you do not want to share your information using NDA. If so, contact the researchers who conducted this study, and they will tell NDA, which can stop sharing the research information. However, NDA cannot take back information that was shared before you changed your mind. If you would like more information about NDA, this is available on-line at http://data-archive.nimh.gov.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### COMPENSATION AND ECONOMIC CONSIDERATIONS

You will not be charged for any procedures that are a part of this study, including the study medication. We offer reasonable compensation for travel costs related to your study participation. You must bring in receipts for these costs, and compensation is limited to no more than \$10 per week.

To compensate you for the time required for each weekly study visit, we offer \$25 at the Week 0, Week 1, Week 2, and Week 3 visit (\$100 total if you attend all visits). This money will be paid by cash at the conclusion of each of these visits.

To compensate you for the time required for the brain scans, we offer \$50 for each MRI scan and \$150 for each PET scan (\$400 total if you attend all visits). This money will be paid in 1 lump sum payment at the end of the study. Payments typically require 1-3 weeks to process and will be mailed in the form of a check.

### RESEARCH STANDARDS

Federal regulations require that we inform participants about our institution's policy with regard to compensation and payment for treatment of research-related injuries.

If you believe that you have sustained an injury as a result of participating in a research study, you may contact the Principal Investigator at 646-774-8660 so that you can review the matter and identify the medical resources that may be available to you.

Please be aware that:

- 1. The New York State Psychiatric Institute, Columbia University and New York Presbyterian Hospital will furnish that emergency medical care determined to be necessary by the medical staff of this hospital
- 2. You will be responsible for the cost of such care, either personally or through your medical insurance or other form of medical coverage.
- 3. No monetary compensation for wages lost as a result of injury will be paid to you by the New York State Psychiatric Institute, Columbia University or by New York Presbyterian Hospital.
- 4. By signing this consent form, you are not waiving any of your legal rights to seek compensation through the courts.

### **QUESTIONS**



If you have further questions about the research procedures, or about your response to the procedures research staff members are available to answer them to the best of their ability. You can reach Dr. Bret Rutherford at 646-774-8660 during general business hours. In an emergency, you may reach the on call doctor at 917-786-6940, 24 hours per day. If you have general questions, you may contact the research coordinator at 646-774-8664. We will notify you of any significant new findings that may relate to your willingness to continue to participate.

If you have any questions about your rights as a research participant, want to provide feedback, or have a complaint, you may call the NYSPI Institutional Review Board (IRB). (An IRB is a committee that protects the rights of human subjects in research studies). You may call the IRB Main Office at (646) 774-7155 during regular office hours.

You will be given a copy of this consent form to keep.

### DOCUMENTATION OF CONSENT

I have read the above and voluntarily agree to participate in the research study described above. To the best of my knowledge, I am not pregnant. I have been informed that my participation is voluntary, and that I can withdraw from the study at any time without penalty or loss of benefits to which I am otherwise entitled.

| Print name: | |
|---|---|
| Signed: | |
| Date: | |
| benefits, and alternatives to particip | ed research with this participant including the risks, pation (including the alternative of not participating in ad an opportunity to ask questions and in my opinion articipate in this research. |
| Print name: | |
| Person Designated to Obtain Conse | ent |
| Signed: | |
| Date: | |